CLINICAL TRIAL: NCT00628173
Title: Results of Different Location of Ahmed Glaucoma Valve Implantation in Refractory Glaucoma, Superior Versus Inferior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8417
Record Dates: First submitted 2008-02-25; First posted 2008-03-04 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-02

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

ARMS (2):
- 1 (Experimental): patients with refractory glaucoma who were candidate for AGV implantation allocated in superior site
  Interventions: Procedure: AGV implantation
- 2 (Experimental): patients with refractory glaucoma who were candidate for AGV implantation allocated in inferior site
  Interventions: Procedure: AGV implantation

INTERVENTIONS:
Procedure: AGV implantation

SUMMARY:
Purpose:To compare the efficacy and safety of Ahmed Glaucoma Valve (AGV) implantation in the superior versus inferior quadrants.

Methods: In a non-randomized clinical trial and over a period of two years, consecutive patients with refractory glaucoma underwent AGV implantation in the superior or inferior quadrants. Main outcome measures included best corrected visual acuity (BCVA), intraocular pressure (IOP), number of glaucoma medications, complications and success rate (defined as at least 30% IOP reduction below preoperative values and 5<IOP<22 mmHg with or without glaucoma medications). Other criteria for failure included implant removal, additional glaucoma surgery, phthisis bulbi or loss of light perception.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory glaucoma who need AGV implantation

Exclusion Criteria:

* Eyes with less than 3 months follow-up
* Severe conjunctival adhesions and scarring for the site of surgery
* Presence of thin sclera and staphyloma for the site of surgery
* The presence or anticipated need for silicone oil for superior implantation
* Active neovascular glaucoma for inferior implantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2005-01; Primary Completion 2007-05; Study Completion 2007-12